CLINICAL TRIAL: NCT01395732
Title: Effects of Bosentan in a Homogenous Population of Systemic Sclerosis Subjects With a Predefined Restriction of Blood Flow in the Hands
Brief Title: Bosentan in Systemic Sclerosis
Acronym: HOME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-052-427
Record Dates: First submitted 2011-07-06; First posted 2011-07-18 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Systemic Sclerosis; Digital Ulcers
MeSH Terms: conditions — Scleroderma, Systemic; digital ulcers | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Bosentan — 2 tablets of 62.5 mg a day from baseline to week 4, then 2 tablets of 125 mg per day to week 12.

SUMMARY:
The effect of bosentan on digital ulcers (DU) was studied in two randomized placebo-controlled trials (RAPIDS-1 and RAPIDS-2). A limitation of these studies was the heterogeneous study population. More importantly, there were no endpoints that assessed changes in vasculopathy and / or perfusion. Laser Doppler imaging has been shown to effectively demonstrate blood flow restrictions in the hands of patients with Systemic Sclerosis (SSc). The relation between blood flow restriction in the hands measured by laser Doppler imaging and the extent of DU disease has not been studied. The current study will attempt to demonstrate this relation. In addition, the impact of bosentan on the blood flow in the hands, in a defined cohort of SSc-DU patients with a history of DU within the past 2 years and a clinically relevant reduction of blood flow in the hands, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects > 18 years diagnosed with SSc;
* Reduction of blood flow measured by laser Doppler imaging, of at least 50%, distally to the proximal interphalangeal joint, compared to the healthy volunteers;
* Women of childbearing potential must have a negative pregnancy test and use a reliable form of contraception;
* A history of 1 or more DUs within 2 years prior to inclusion;
* No use of bosentan in the past;
* Subjects willing and able to sign informed consent.

Exclusion Criteria:

* Parenteral prostanoid treatment for DU < 3 months ago;
* Chronic treatment with PDE-5 inhibitor or ERA;
* History of bosentan use
* Irreversible significant limitation of the hand function, e.g. amputation of more than one finger;
* Other types of system- or connective tissue diseases;
* Significant peripheral (macro-) vascular disease due to e.g. diabetes, hyperlipidemia, uncontrolled systemic hypertension, coagulopathy;
* Any serious medical co morbidity (eg, active malignancy) such that the subjects life expectancy is < 12 months;
* Known AST and/or ALT elevations higher than 3 times Upper Limit Normal (ULN);
* Moderate to severe liver function disorder;
* Pregnancy or breastfeeding;
* Treatment with Glibenclamide, Fluconazole, Cyclosporin A, Tacrolimus or other calcineurin inhibitors;
* Hypersensitivity for bosentan or one of its components;
* Subjects not able to follow the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Mean blood flow restriction in patients | Baseline to 12 weeks
  Relationship between blood flow in the hands, as measured by laser Doppler imaging, and extent of Digital Ulcer disease assessed by the mean blood flow restriction in four distinct groups of patients: patients without current Digital Ulcers (pitting scars allowed), patients with new Digital Ulcers (< 3 months), patients with persistent Digital Ulcers (> 3 months) and patients with significant tip-necrosis.

SECONDARY OUTCOMES:
Change in blood flow in the hands | Baseline to 12 weeks of bosentan treatment
  Change in blood flow in the hands after 12 weeks of bosentan treatment compared to the baseline, as measured by laser Doppler imaging.